CLINICAL TRIAL: NCT05101265
Title: An Open-Label, Multicenter, Pharmacokinetic Study of Lurbinectedin in Patients With Advanced Solid Tumors and Varying Degrees of Hepatic Impairment
Brief Title: Clinical Pharmacokinetic Study of Lurbinectedin in Patients With Advanced Solid Tumors and Varying Degrees of Hepatic Impairment
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM1183-A-017-20; 2020-002789-14 (EudraCT Number)
Record Dates: First submitted 2021-09-29; First posted 2021-11-01 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Advanced Solid Tumor; Hepatic Impairment
Keywords: Hepatic Impairment; Advanced Solid Tumor; Lurbinectedin
MeSH Terms: interventions — PM 01183

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, parallel, phase Ib, hepatic impairment study in patients with advanced solid tumors who either have HI at varying degrees (mild, moderate or severe) or qualify for the control group (normal hepatic function) according to the National Cancer Institute Organ Dysfunction Working Group (NCI-ODWG) classification criteria of HI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Normal Hepatic function cohort (Experimental): Patients in the control cohort must meet the following criteria:
  * Total bilirubin ≤ 1.0 x upper limit of normal (ULN) and no clinical (or histological) evidence of liver disease.
  * Aspartate aminotransferase (AST) ≤ 1.0 x ULN and alanine aminotransferase (ALT) ≤ 1.0 x ULN.
  * Albumin ≥ 3.5 g/dL.
  * The age, weight and CLcr should be within ±10 years, ±15 kg and ±20 mL/min of the mean of pooled HI cohort, respectively; and with a similar male/female ratio.
  Interventions: Drug: Lurbinectedin
- Mild Hepatic impairment cohort (Experimental): Patients with Mild Hepatic impairment must meet the following additional criteria
  * Total bilirubin ≤ 1.0 x ULN and AST > 1.0 x ULN, or
  * Total bilirubin > 1.0 - ≤ 1.5 x ULN and any AST, and
  * Albumin ≥ 3.0 g/dL
  Interventions: Drug: Lurbinectedin
- Moderate Hepatic impairment cohort (Experimental): Patients with Moderate Hepatic impairment must meet the following additional criteria
  * Total bilirubin >1.5 - ≤ 3.0 x ULN and any AST, and
  * Albumin ≥ 2.8 g/dL
  Interventions: Drug: Lurbinectedin
- Severe Hepatic impairment cohort (Experimental): Patients with Severe Hepatic impairment must meet the following additional criteria:
  * Total bilirubin >3.0 x ULN and any AST, and
  * Albumin ≥ 2.5 g/dL
  Interventions: Drug: Lurbinectedin

INTERVENTIONS:
Drug: Lurbinectedin — Patients will receive lurbinectedin as a 1-hour (-5/+20 min) i.v. infusion on Day 1 every three weeks (q3wk), over a minimum of 100 mL dilution on 5% glucose or 0.9% sodium chloride via a central line (or a minimum of 250 mL dilution if a peripheral line is used). Of note, Cycle 2 or subsequent will be administered every q3wk (+ 48 hours). Patients will receive a maximum of two cycles: a first mandatory cycle with all study assessments followed by a second optional cycle with lurbinectedin (this last optional for patients with clinical benefit as per Investigator's criteria).
  After completing Cycle 2, those patients waiting for the compassionate use approval will continue on the study receiving lurbinectedin herein after until disease progression, unacceptable toxicity, consent withdrawal or while it is considered to be in their best interest, or until starting treatment with lurbinectedin under a Compassionate Use Agreement outside this study.
  Lurbinectedin at a 3.2 mg/m² dose.
  Other Names: PM1183
  Arms: Mild Hepatic impairment cohort; Normal Hepatic function cohort
Drug: Lurbinectedin — Patients will receive lurbinectedin as a 1-hour (-5/+20 min) i.v. infusion on Day 1 every three weeks (q3wk), over a minimum of 100 mL dilution on 5% glucose or 0.9% sodium chloride via a central line (or a minimum of 250 mL dilution if a peripheral line is used). Of note, Cycle 2 or subsequent will be administered every q3wk (+ 48 hours). Patients will receive a maximum of two cycles: a first mandatory cycle with all study assessments followed by a second optional cycle with lurbinectedin (this last optional for patients with clinical benefit as per Investigator's criteria).
  After completing Cycle 2, those patients waiting for the compassionate use approval will continue on the study receiving lurbinectedin herein after until disease progression, unacceptable toxicity, consent withdrawal or while it is considered to be in their best interest, or until starting treatment with lurbinectedin under a Compassionate Use Agreement outside this study.
  Lurbinectedin at a 1.6 mg/m² dose
  Other Names: PM1183
  Arms: Moderate Hepatic impairment cohort; Severe Hepatic impairment cohort

SUMMARY:
Lurbinectedin is mainly eliminated by the liver. Thus, Hepatic Impairment (HI) may alter the plasma concentrations of lurbinectedin. This study is designed to examine the PK and safety of an adjusted dose of lurbinectedin when administered to patients with HI. The results of this study may be used to support future clinical studies in patients and prescribing information in future labeling.

DETAILED DESCRIPTION:
This is a prospective, open-label, parallel, phase Ib, hepatic impairment study in patients with advanced solid tumors who either have Hepatic Impairment (HI) at varying degrees (mild, moderate or severe) or qualify for the control group (normal hepatic function) according to the National Cancer Institute Organ Dysfunction Working Group (NCI-ODWG) classification criteria of HI.

ELIGIBILITY:
Inclusion criteria

All patients must fulfill the following inclusion criteria (1 - 9) to be enrolled in the study:

1. Voluntary signed and dated written informed consent prior to any specific study procedure.
2. Male or female with age ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2.
4. Life expectancy > 1 month.
5. Pathologically confirmed diagnosis of advanced solid tumors [except for primary central nervous system (CNS) tumors], for which no standard therapy exists.
6. Recovery to grade ≤ 1 from drug-related adverse events (AEs) of previous treatments, excluding alopecia and/or cutaneous toxicity and/or peripheral neuropathy and/or fatigue grade ≤ 2, according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCICTCAE v.5).
7. Laboratory values within fourteen days prior to registration:

   1. Absolute neutrophil count (ANC) > 2.0 x 10^9/L, platelet count > 120 x 10^9/L and hemoglobin > 9.0 g/dL (patients may be transfused as clinically indicated prior to study entry).
   2. Creatinine clearance (CLcr) ≥ 30 mL/min (using Cockcroft and Gault's formula).
   3. Creatine phosphokinase (CPK) ≤ 2.5 x ULN (≤ 5.0 x ULN if disease related).
8. Evidence of non-childbearing status for women of childbearing potential
9. History of alcohol abuse is permissible providing that the results of alcohol (in breath or blood) test are negative at screening.

   Patients in the control cohort (normal hepatic function) must meet the following additional inclusion criteria (10 - 13) to be enrolled in the study:
10. Total bilirubin ≤ 1.0 x upper limit of normal (ULN) and no clinical (or histological) evidence of liver disease.
11. Aspartate aminotransferase (AST) ≤ 1.0 x ULN and alanine aminotransferase (ALT) ≤ 1.0 x ULN.
12. Albumin ≥ 3.5 g/dL.
13. The age, weight and CLcr should be within ±10 years, ±15 kg and ±20 mL/min of the mean of pooled HI cohort, respectively; and with a similar male/female ratio.

    Patients with HI must meet the following additional inclusion criteria (14 - 16):
14. Patients with HI per cohort must meet:

    a) Mild HI cohort:

    i) Total bilirubin ≤ 1.0 x ULN and AST > 1.0 x ULN, or

    ii) Total bilirubin > 1.0 - ≤ 1.5 x ULN and any AST, and

    iii) Albumin ≥ 3.0 g/dL

    b) Moderate HI cohort:

    i) Total bilirubin >1.5 - ≤ 3.0 x ULN and any AST, and

    ii) Albumin ≥ 2.8 g/dL

    c) Severe HI cohort:

    i) Total bilirubin >3.0 x ULN and any AST, and

    ii) Albumin ≥ 2.5 g/dL
15. Documented liver disease and/or hepatic metastases, with physical examination, liver biopsy or hepatic ultrasound, CT scan or MRI consistent with diagnosis.
16. Stable HI, defined as no clinically significant change in the disease status within the last 14 days, as documented by the patient's recent medical history (e.g., no worsening clinical signs of HI, or no worsening of total bilirubin or prothrombin time by more than 50%).

Exclusion criteria

All patients who meet any of the following criteria (1 - 6) will be excluded from participating in the study:

1. Concomitant diseases/conditions:

   1. History or presence of unstable angina, myocardial infarction, congestive heart failure, or clinically significant valvular disease within last year.
   2. Symptomatic arrhythmia or any uncontrolled arrhythmia.
   3. Active infection by hepatitis B virus (HBV) or hepatitis C virus (HCV), defined as: for hepatitis B, positive test for quantitative Hepatitis B virus polymerase chain reaction (PCR or HBV-DNA+), regardless of the HBsAg; and for hepatitis C, positive test for quantitative Hepatitis C virus by PCR (or HCV-RNA+).
   4. Human immunodeficiency virus (HIV)-positive patients.
   5. History of Gilbert's syndrome diagnosis.
   6. History of biliary sepsis in the past 2 months.
   7. Patients with biliary obstruction for which a stent has been placed are eligible, provided the stent has been in place for at least 10 days prior to the first dose of lurbinectedin and the liver function has stabilized; two measurements at least 2 days apart that put the patient in the same hepatic dysfunction cohort will be accepted as evidence of stable hepatic function; there should be no evidence of biliary sepsis.
   8. Active coronavirus disease of 2019 (COVID-19) disease (this includes positive test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in nasopharyngeal/oropharyngeal swabs or nasal swabs by PCR).
2. Symptomatic, progressive or corticosteroids-requiring documented brain metastases or leptomeningeal disease involvement. Patients with asymptomatic documented stable brain metastases not requiring corticosteroids during the last four weeks are allowed.
3. Use of (strong or moderate) inhibitors or inducers of CYP3A4 activity within three weeks prior to Day 1 of Cycle 1.
4. Less than three weeks since the last systemic anticancer therapy (investigational or standard), or less than two weeks since last radiotherapy before starting treatment of Day 1 of Cycle 1. Treatment with any other investigational product within the 30 days before Day 1 of Cycle 1.
5. Women who are pregnant or breast-feeding and fertile patients (men and women) who are not using an effective method of contraception.
6. Psychiatric illness/social situations that would limit compliance with study requirements.

   Patients with HI (all cohorts) who meet any of the following additional criteria (7 - 9) will be excluded:
7. History of gastrointestinal hemorrhage due to esophageal varices or peptic ulcers less than one month prior to Day 1 of Cycle 1.
8. Signs of significant hepatic encephalopathy (> grade II Portal Systemic Encephalopathy).
9. Severe ascites and/or pleural effusion, except for patients at the severe HI cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Total plasma dose-normalized Cmax | Preinfusion, 5 minutes before end of infusion, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, 96 hours, 168 hours, 240 hours, 336 hours, and 504 hours after end of infusion
  Total plasma dose-normalized Cmax of lurbinectedin will be compared between Control (normal hepatic function) cohort and each of the Hepatic impairment cohorts
Total plasma dose-normalized AUC0-48h | Preinfusion, 5 minutes before end of infusion, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, 96 hours, 168 hours, 240 hours, 336 hours, and 504 hours after end of infusion
  Total plasma dose-normalized area under curve (AUC) 0-48h of lurbinectedin will be compared between Control (normal hepatic function) cohort and each of the Hepatic impairment cohorts
Total plasma dose-normalized AUC0-∞ | Preinfusion, 5 minutes before end of infusion, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, 96 hours, 168 hours, 240 hours, 336 hours, and 504 hours after end of infusion
  Total plasma dose-normalized AUC0-∞ (if data do not permit so, AUC0-t will be used) of lurbinectedin will be compared between Control (normal hepatic function) cohort and each of the Hepatic impairment cohorts

SECONDARY OUTCOMES:
Total plasma dose-normalized AUC0-t | Preinfusion, 5 minutes before end of infusion, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, 96 hours, 168 hours, 240 hours, 336 hours, and 504 hours after end of infusion
  Change in dose-normalized total AUC0-t of lurbinectedin between Control (normal hepatic function) cohort and each of the Hepatic impairment cohorts will be explored.
Clearance | Preinfusion, 5 minutes before end of infusion, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, 96 hours, 168 hours, 240 hours, 336 hours, and 504 hours after end of infusion
  Change in Clearance (Cl) of lurbinectedin between Control (normal hepatic function) cohort and each of the Hepatic impairment cohorts will be explored.
Volume of Distribution at Steady State | Preinfusion, 5 minutes before end of infusion, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, 96 hours, 168 hours, 240 hours, 336 hours, and 504 hours after end of infusion
  Change in Volume of Distribution at Steady State (Vss) of lurbinectedin between Control (normal hepatic function) cohort and each of the Hepatic impairment cohorts will be explored.
T1/2 | Preinfusion, 5 minutes before end of infusion, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, 96 hours, 168 hours, 240 hours, 336 hours, and 504 hours after end of infusion
  Change in T1/2 of lurbinectedin between Control (normal hepatic function) cohort and each of the Hepatic impairment cohorts will be explored.
Dose-normalized unbound AUCu,0-∞ | Preinfusion, 5 minutes before end of infusion, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, 96 hours, 168 hours, 240 hours, 336 hours, and 504 hours after end of infusion
  Change in dose-normalized unbound AUCu,0-∞ of lurbinectedin between Control (normal hepatic function) cohort and each of the Hepatic impairment cohorts will be explored.
Dose-normalized unbound AUCu,0-48h | Preinfusion, 5 minutes before end of infusion, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, 96 hours, 168 hours, 240 hours, 336 hours, and 504 hours after end of infusion
  Change in dose-normalized unbound AUCu,0-48h of lurbinectedin between Control (normal hepatic function) cohort and each of the Hepatic impairment cohorts will be explored.
Dose-normalized unbound AUCu,0-t | Preinfusion, 5 minutes before end of infusion, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, 96 hours, 168 hours, 240 hours, 336 hours, and 504 hours after end of infusion
  Change in dose-normalized unbound AUCu,0-t of lurbinectedin between Control (normal hepatic function) cohort and each of the Hepatic impairment cohorts will be explored.
Dose-normalized unbound Cu,max | Preinfusion, 5 minutes before end of infusion, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, 96 hours, 168 hours, 240 hours, 336 hours, and 504 hours after end of infusion
  Change in dose-normalized unbound Cu,max of lurbinectedin between Control (normal hepatic function) cohort and each of the HI cohorts will be explored.
Unbound CLu | Preinfusion, 5 minutes before end of infusion, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, 96 hours, 168 hours, 240 hours, 336 hours, and 504 hours after end of infusion
  Change in CLu of lurbinectedin between Control (normal hepatic function) cohort and each of the Hepatic impairment cohorts will be explored.
Unbound Vss,u | Preinfusion, 5 minutes before end of infusion, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, 96 hours, 168 hours, 240 hours, 336 hours, and 504 hours after end of infusion
  Change in Vss,u of lurbinectedin between Control (normal hepatic function) cohort and each of the Hepatic impairment cohorts will be explored.
T1/2,u | Preinfusion, 5 minutes before end of infusion, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, 96 hours, 168 hours, 240 hours, 336 hours, and 504 hours after end of infusion
  Change in T1/2,u of lurbinectedin between Control (normal hepatic function) cohort and each of the Hepatic impairment cohorts will be explored.
Ratios total AUC0-∞ | Preinfusion, 5 minutes before end of infusion, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, 96 hours, 168 hours, 240 hours, 336 hours, and 504 hours after end of infusion
  Change in ratios between total AUC0-∞ of main lurbinectedin metabolites relative to parent drug between Control (normal hepatic function) cohort and each of the Hepatic impairment cohorts will be explored.
Ratios AUC0-48h | Preinfusion, 5 minutes before end of infusion, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, 96 hours, 168 hours, 240 hours, 336 hours, and 504 hours after end of infusion
  Change in ratios between total AUC0-48h of main lurbinectedin metabolites relative to parent drug between Control (normal hepatic function) cohort and each of the Hepatic impairment cohorts will be explored.
Ratios AUC0-t | Preinfusion, 5 minutes before end of infusion, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, 96 hours, 168 hours, 240 hours, 336 hours, and 504 hours after end of infusion
  Change in ratios between total AUC0-t of main lurbinectedin metabolites relative to parent drug between Control (normal hepatic function) cohort and each of the Hepatic impairment cohorts will be explored.
Ratios Cmax | Preinfusion, 5 minutes before end of infusion, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 24 hours, 48 hours, 96 hours, 168 hours, 240 hours, 336 hours, and 504 hours after end of infusion
  Change in ratios between total Cmax of main lurbinectedin metabolites relative to parent drug between Control (normal hepatic function) cohort and each of the Hepatic impairment cohorts will be explored.
Percentage of patients with non-serious adverse events | From first infusion to the end-of-treatment visit which will be scheduled within 31 days (±10 days) after administration of the last dose of lurbinectedin
  Treatment safety (AEs) will be graded according to the NCI-CTCAE v.5.
Percentage of patients with serious adverse events | From first infusion to the end-of-treatment visit which will be scheduled within 31 days (±10 days) after administration of the last dose of lurbinectedin
  Treatment safety (SAEs) will be graded according to the NCI-CTCAE v.5.
Percentage of patients with Laboratory abnormalities | From first infusion to the end-of-treatment visit which will be scheduled within 31 days (±10 days) after administration of the last dose of lurbinectedin
  Laboratory abnormalities will be graded according to the NCI-CTCAE v.5.
Pharmacogenetics | After first cycle (21 days)
  The presence or absence of PGt polymorphisms in genes relevant for lurbinectedin disposition (distribution, metabolism and excretion) from a single blood sample collected at any time during the trial (but preferably at the same time as the pre-treatments PK sample on Day 1 of Cycle 1), which will be stored to explain individual variability in main PK parameters in future analyses

CONTACTS AND LOCATIONS:
Overall Officials: Rubin Lubomirov, MD, PhD, Study Director — PharmaMar; Sara Martínez González, MD, Study Director — PharmaMar
Locations (6):
- Spain (6):
  - Hospital Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Universitari Vall d'Hebron, Barcelona, Catalonia
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jimenez Diaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid